CLINICAL TRIAL: NCT07354685
Title: The Effect of a Psychological Resilience Program for Phubbing on Nursing Students' Communication Skills and Phubbing Behaviors: A Randomized Controlled Trial
Brief Title: The Effect of the Developed Psychological Resilience Program on Phubbing Behaviors and Communication Skills
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Mert Hızlıoğluları, PhD Candidate, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ETK00-2025-0132
Record Dates: First submitted 2026-01-05; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Phubbing
Keywords: Phubbing; Nursing Students; Communication Skills; psychological resilience

STUDY DESIGN:
Intervention Model Description: The intervention in this study consists of a structured psychological resilience development program comprising eight modules. The program is designed to support nursing students in coping more effectively with academic, social, and interpersonal challenges encountered during university life. The modules include activities aimed at enhancing self-awareness, emotional strength, healthy communication, stress management, and interpersonal skills. The program is delivered in a group-based format, with each module planned to build upon and complement the others.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Psychological Resilience-Based Sociotelism Prevention Program (Experimental): Intervention Arm:
  Psychological Resilience Development Program for Phubbing
  Interventions: Behavioral: Psychological Resilience Development Program for Phubbing
- Control Arm (No Intervention): Control Arm

INTERVENTIONS:
Behavioral: Psychological Resilience Development Program for Phubbing — This study evaluates the effectiveness of an 8-module psychological resilience development program designed to address phubbing behaviors among participants. The program was structured to enhance individuals' capacity to cope with digital distractions and strengthen adaptive psychosocial skills in interpersonal contexts. The intervention aims to improve communication skills, increase psychological resilience levels, and reduce sociotelism tendencies by promoting mindful technology use, emotional regulation, and awareness of face-to-face interaction dynamics. The impact of the program is assessed through pre- and post-intervention measurements, allowing for a systematic examination of changes in participants' communication competencies, resilience capacities, and sociotelism levels following completion of the eight modules.
  Arms: Intervention Arm: Psychological Resilience-Based Sociotelism Prevention Program

SUMMARY:
The goal of this study is to determine whether a psychological resilience-based intervention program developed to prevent sociotelism is effective in nursing students. The study also aims to evaluate the feasibility and acceptability of the program.

The main questions this study aims to answer are:

Does the psychological resilience development program reduce sociotelism behaviors among nursing students?

Does the program improve nursing students' communication skills?

Researchers will compare nursing students who participate in the psychological resilience development program with those in a control group who do not receive the intervention, in order to determine whether the program is effective in reducing sociotelism behaviors and enhancing communication skills.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate nursing students aged 18 - 30 years old
* Voluntary participation
* Ability to understand and complete self-report questionnaires.

Exclusion Criteria:

* Presence of a diagnosed severe psychiatric disorder
* Current participation in another psychological intervention program.

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Communication Skills Level | Baseline (pre-intervention) and immediately after the 8-module intervention (post-intervention)
  The Communication Skills Scale was developed by Fidan Korkut Owen and Aslı Bugay in 2014. The scale consists of 25 items organized into four subdimensions. Higher scores indicate higher levels of communication skills. For both the total scale and its subdimensions, mean item total scores are used.
  The scale is a 5-point Likert-type instrument, rated as follows:
  (1 = Never, 2 = Rarely, 3 = Occasionally, 4 = Often, 5 = Always).
  The Cronbach's alpha coefficient for the Communication Skills Scale was found to be 0.88, indicating high internal consistency. Total scores range from 25 to 125, with higher scores reflecting more advanced communication skills
  The four subdimensions of the scale and their corresponding item numbers are as follows:
  1. Communication Relationships and Basic Skills
  2. Self-Expression
  3. Active Listening and Nonverbal Communication
  4. Willingness to Communicate
Psychological Resilience Level | Baseline (pre-intervention) Immediately after the 8-module intervention (post-intervention)
  Psychological resilience will be assessed using the Psychological Resilience Scale for Adults. The scale consists of 33 items rated on a 5-point Likert scale (1 = Never to 5 = Always). Total scores range from 33 to 165, with higher scores indicating greater psychological resilience.
Levels of Phubbing Behavior and Exposure to Phubbing Level | Baseline (pre-intervention) and immediately after the 8-module intervention (post-intervention)
  In this study, the Phubbing Behaviors Scale was used as the data collection instrument. The scale was originally developed by Chotpitayasunondh and Douglas (2018) and was adapted into Turkish by Derya Orhan Göksun (2019), who conducted its validity and reliability analyses. The scale consists of two sections and is rated on a 7-point Likert scale.
  The first section is the Generic Scale of Phubbing (GSP), which consists of 15 items grouped into four subdimensions. The Cronbach's alpha coefficient for this section was 0.78. Total scores range from 15 to 105, calculated by summing the Likert-scale responses provided by the participants. All items in this section are negatively worded within the context of social norms and general acceptance; therefore, higher total scores indicate more negative outcomes, reflecting higher levels of phubbing behavior. In summary, as the total score increases, the the level of phubbing behavior also increases.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical restrictions, confidentiality considerations, and the protection of participants' privacy in accordance with ethical approval and informed consent.